CLINICAL TRIAL: NCT06297083
Title: Analysing HIgh Dose Probiotic Peanut Oral Immunotherapy (PPOIT) and High Dose Peanut Oral Immunotherapy (OIT) Versus LOw Dose Peanut OIT for Peanut Allergy
Acronym: HILO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Delays in manufacturing & increased costs of materials, manufacturing and logistics identified during trial set up caused the trial budget to exceed the available funds and an inability to complete the study within required grant timelines.
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 100992 HILO
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Intervention Model Description: This is a three-arm, multi-center, head-to-head randomized study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, outcome assessors, other research staff, treating clinicians, investigators and trial statistician will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- High-dose peanut OIT combined with probiotic (HD PPOIT) (Experimental): High-dose rapid escalation peanut OIT combined with probiotic (HD PPOIT) taken daily for 18 months.
  Interventions: Drug: Peanut Oral Powder [PEANUT POWDER]; Dietary Supplement: Probiotic (LGG®, Lactobacillus Rhamnosus) or placebo probiotic (maltodextrin)
- High-dose peanut OIT combined with probiotic placebo (HD OIT) (Experimental): High-dose rapid escalation peanut OIT combined with probiotic placebo (HD OIT) taken daily for 18 months
  Interventions: Drug: Peanut Oral Powder [PEANUT POWDER]; Dietary Supplement: Probiotic (LGG®, Lactobacillus Rhamnosus) or placebo probiotic (maltodextrin)
- Low-dose peanut OIT combined with probiotic placebo (LD OIT) (Active Comparator): Low-dose slow escalation peanut OIT combined with probiotic placebo (LD OIT) taken daily for 18 months.
  Interventions: Drug: Peanut Oral Powder [PEANUT POWDER]; Dietary Supplement: Probiotic (LGG®, Lactobacillus Rhamnosus) or placebo probiotic (maltodextrin)

INTERVENTIONS:
Drug: Peanut Oral Powder [PEANUT POWDER] — Peanut oral immunotherapy at varying doses and build-up regimes given daily for 18 months
  Other Names: Peanut oral immunotherapy
Dietary Supplement: Probiotic (LGG®, Lactobacillus Rhamnosus) or placebo probiotic (maltodextrin) — Probiotic or placebo-probiotic given daily for 18 months

SUMMARY:
This study will compare the effectiveness of three different treatments to treat peanut allergy

DETAILED DESCRIPTION:
This is a three-arm, multi-centre, head-to-head randomised trial, comparing two treatments against a low dose oral immunotherapy approach for peanut allergy.

One hundred and thirty children aged 1 year to 10 years with current peanut allergy confirmed by failed double-blind placebo-controlled food challenge (DBPCFC) at study screening will be recruited for this study. Participants will be recruited from The Royal Children's Hospital Melbourne, Women's and Children's Hospital (Adelaide) and from the general community.

Participants will be randomized to:

1. High-dose rapid escalation peanut OIT combined with probiotic (HD PPOIT)
2. High-dose rapid escalation peanut OIT combined with probiotic placebo (HD OIT)
3. Low-dose slow escalation peanut OIT combined with probiotic placebo (LD OIT)

The length of the treatment period for each participant is 18 months and the post-treatment follow up period is 12 months

ELIGIBILITY:
Inclusion Criteria:

* Aged 1-10 years.
* >7kg (the weight considered safe for the administration of an adrenaline injector);
* Confirmed diagnosis of peanut allergy as defined by a failed DBPCFC with peanut and a positive SPT or sIgE to peanut at screening;
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf

Exclusion Criteria:

* History of severe anaphylaxis (as defined by persistent hypotension, collapse, loss of consciousness, persistent hypoxia or ever needing more than three (3) doses of intramuscular adrenaline or an intravenous adrenaline infusion for management of an allergic reaction)
* Severe anaphylaxis during the study entry DBPCFC (defined as persistent hypotension, collapse, loss of consciousness, persistent hypoxia, or requiring more than 3 doses of intramuscular adrenaline or an intravenous adrenaline infusion for management of an allergic reaction)
* Ongoing chronic persistent asthma (as per Australian Asthma Foundation guidelines)
* Underlying medical conditions (e.g. cardiac disease) that increase the risks associated with anaphylaxis
* Use of beta-blockers, and angiotensin converting enzyme (ACE) inhibitors
* Reacting to the placebo component during the study entry DBPCFC
* Have received other food immunotherapy treatment in the preceding 12 months
* Currently taking immunomodulatory therapy (including allergen immunotherapy)
* Past or current major illness that in the opinion of the Site Investigator may affect the subject's ability to participate in the study e.g. increased risk to the participant
* History of suspected or biopsy-confirmed eosinophilic oesophagitis (EoE)
* Subjects who in the opinion of the Site Investigator are unable to follow the protocol
* Another family member already enrolled in the trial (to maintain blinding, safety and equity of access) or in any other clinical trial from the same study group.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Difference between the treatment arms in the proportion of participants who achieve remission of peanut allergy at 8 weeks post treatment. | 22 months
  Remission will be assessed 8 weeks after the end of treatment timepoint and is defined as passing (completing without reaction) the double-blind placebo controlled food challenge (DBPCFC) at the end of treatment and at 8 weeks post treatment

SECONDARY OUTCOMES:
Difference between the treatment arms in the proportion of participants who achieve full desensitisation of peanut allergy at end of treatment | 20 months
  Full desensitisation will be defined by participants passing (completing without reaction) the double-blind placebo controlled food challenge (DBPCFC) undertaken at the end of treatment
Difference between the treatment arms in the exposure-adjusted event rate of adverse events (AE) | 20 months
  The total number of treatment-related AE the participant reports during the course of treatment adjusted for the time the participant is on treatment (in years)
Difference between treatment arms in changes in Quality of Life Scores using the Food Allergy Quality of Life Questionnaires (FAQLQ). | Baseline, 22weeks, 76 weeks, 84 weeks, 128 weeks
  FAQLQ total score, as well as three sub-scores (food anxiety, general emotional impact, and social and dietary limitations) will be calculated as per the instrument scoring manual
Difference between treatment arms in changes in the peanut skin prick test (SPT) wheal size. | Baseline, 76 weeks, 84 weeks,128 weeks
  Skin prick test to whole peanut extract
Difference between treatment arms in change from baseline peanut specific immunoglobulin E (sIgE) levels | Baseline, 76 weeks, 84 weeks,128 weeks
  Blood samples will be collected and levels of sIgE against peanut will be measured by ImmunoCAP (Phadia AB, Uppsala, Sweden)
Difference between treatment arms in adherence to treatment regime as measured by daily treatment doses taken by the participant | 20 months
  Adherence to treatment will be monitored by reviewing the participant diary
Difference between treatment arms in participant experience as assessed from qualitative interviews | 20 months
  Interview guide developed and conducted, recorded, transcribed verbatim, and responses explored using framework analysis
Difference between clinical outcome groups in cost using the Consolidated Health Economic Evaluation Reporting Standards (CHEERS) | Baseline through to 32 months
  Captured per number of hospitalizations, Emergency room (ER) visits, General Practitioner (GP) visits and medications / number of prescriptions required. Data acquired using participant questionnaires, participant study diaries and supplemented by administrative hospital data linkage
Difference between clinical outcome groups in quality adjusted life year (QALY) will be estimated at 32 months using the Food Allergy Quality of Life Form (FAQLQ) mapped to the generic health utility instrument Assessment of Quality of Life-6D (AQoL-6D) | 32 months
Difference between clinical outcome groups in peanut ingestion from end of treatment to 12 months post treatment | 20 months to 32 months
  Peanut ingestion data will be captured from the participant's study diary
Difference between clinical outcome groups in reactions to peanut from end of treatment to 12 months post treatment | 20 months to 32 months
  Number of reactions, symptoms experienced, and treatment administered will be captured from the participant's study diary

CONTACTS AND LOCATIONS:
Overall Officials: Paxton Loke, Principal Investigator — Murdoch Childrens Research Institute

IPD SHARING:
Plan to Share IPD: Yes
Beginning 24 months after article publication, the following will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access (including any conditions relating to MCRI's intellectual property):
  * Individual participant data that underlie the results reported in this article after de-identification (text, tables, figures and appendices)
  * Trial protocol, Statistical Analysis Plan, Informed Consent Form (ICF)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 24 months following article publication
Access Criteria: These will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access (including any conditions relating to MCRI's intellectual property)
URL: https://www.melbournechildrens.com/mctc/

REFERENCES:
- [Background] Loke P, Orsini F, Lozinsky AC, Gold M, O'Sullivan MD, Quinn P, Lloyd M, Ashley SE, Pitkin S, Axelrad C, Metcalfe JR, Su EL, Tey D, Robinson MN, Allen KJ, Prescott SL, Galvin AD, Tang MLK; PPOIT-003 study group. Probiotic peanut oral immunotherapy versus oral immunotherapy and placebo in children with peanut allergy in Australia (PPOIT-003): a multicentre, randomised, phase 2b trial. Lancet Child Adolesc Health. 2022 Mar;6(3):171-184. doi: 10.1016/S2352-4642(22)00006-2. Epub 2022 Feb 4. PMID 35123664